CLINICAL TRIAL: NCT00764400
Title: Communication Outcomes for Naming Treatments in Aphasia
Brief Title: Treatment for Word Retrieval Impairments in Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Dr. Anastasia Raymer, Professor of Communications Disorders & Special Education, Old Dominion University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R15DC009690 (NIH); 3R15DC009690 (NIH)
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Stroke
Keywords: aphasia; anomia; speech therapy; rehabilitation
MeSH Terms: conditions — Stroke; Aphasia; Anomia; Communication Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Errorless Naming Treatment (Experimental)
  Interventions: Behavioral: Word Retrieval Treatments for Aphasia
- Verbal+Gestural Facilitation (Experimental)
  Interventions: Behavioral: Word Retrieval Treatments for Aphasia

INTERVENTIONS:
Behavioral: Word Retrieval Treatments for Aphasia — Speech therapy sessions take place 4 times per week for up to 90 minutes per session. Following a phase of baseline pre-testing, two phases of speech therapy will take place lasting up to 20 sessions per phase. Post-testing will take place immediately upon completion of the treatment phases and again at 1 month post study completion.

SUMMARY:
In this study the investigators are examining the effectiveness of two different speech therapy protocols for word retrieval impairments experienced by individuals with stroke-induced aphasia. One treatment involves errorless naming treatment and the other employs verbal plus gestural facilitation of word retrieval. Participants will receive one of the two treatments over several months. Before and after treatment the investigators will administer several tests and conversational samples to examine changes associated with the treatments. The investigators hypothesize that, whereas both treatments will lead to improvements in words rehearsed in therapy, communication outcomes in conversation will be broader for the verbal plus gestural protocol.

DETAILED DESCRIPTION:
In this study the investigators are examining the effectiveness of two different speech therapy protocols for word retrieval impairments experienced by individuals with stroke-induced aphasia. One treatment involves errorless naming treatment and the other employs verbal plus gestural facilitation of word retrieval. Participants will receive one of the two treatments over several months. Before and after treatment the investigators will administer several tests and conversational samples to examine changes associated with the treatments. The investigators hypothesize that, whereas both treatments will lead to improvements in words rehearsed in therapy, communication outcomes in conversation will be broader for the verbal plus gestural protocol.

ELIGIBILITY:
Inclusion Criteria:

* left hemisphere stroke >4 months earlier
* aphasia with word retrieval impairments
* >21 years of age right handed
* speaker of English as the preferred language
* >6 grade education

Exclusion Criteria:

* history of developmental learning difficulties
* history of prior neurological illnesses
* chronic medical illnesses that restrict participation in speech therapy
* alcohol or drug dependence
* severe uncorrected impairments of vision or hearing

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-08; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Daily Probe Picture Naming | daily probes from three times per week for up to 3 months and one month posttreatment

SECONDARY OUTCOMES:
Western Aphasia Battery | pre-treatment and at treatment completion
Boston Naming Test | pretreatment and at treatment completion
Discourse Sample | pre-treatment and at treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia M Raymer, PhD, Principal Investigator — Old Dominion University
Locations (1):
- Old Dominion University Speech and Hearing Clinic, Norfolk, Virginia, United States